CLINICAL TRIAL: NCT02351726
Title: Mitroflow Aortic Pericardial Heart Valve With Phospholipid Reduction Treatment Post Approval Study
Brief Title: Mitroflow DL Post Approval Study- North America
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor business decision
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMT001
Record Dates: First submitted 2015-01-22; First posted 2015-01-30 (Estimated); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Aortic Stenosis; Aortic Regurgitation; Aortic Valve Insufficiency; Heart Valve Diseases; Cardiovascular Abnormalities; Cardiovascular Diseases; Congenital Abnormalities; Heart Diseases; Pathological Conditions, Anatomical
Keywords: aortic valve replacement; aortic stenosis; aortic steno-insufficiency
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency; Heart Valve Diseases; Cardiovascular Abnormalities; Cardiovascular Diseases; Congenital Abnormalities; Heart Diseases; Pathological Conditions, Anatomical

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mitroflow DL (Experimental): Treatment with Mitroflow Pericardial Aortic Heart Valve with Phospholipid Reduction Therapy (Model DL)
  Interventions: Device: Mitroflow DL

INTERVENTIONS:
Device: Mitroflow DL — Treatment with Mitroflow Pericardial Aortic Heart Valve with Phospholipid Reduction Therapy (Model DL)
  Other Names: Mitroflow Pericardial Aortic Heart Valve with PRT

SUMMARY:
Prospective, non-randomized, multicenter post-approval study to collect long term clinical and echographic data on Mitroflow DL patients.

DETAILED DESCRIPTION:
The purpose of this clinical investigation is to evaluate the safety and efficacy of the Mitroflow DL valve when used to replace diseased or dysfunctional native or prosthetic aortic heart valves. The study will be conducted in a minimum of 15 centers in the United States. Patients will be evaluated at each of the following time intervals:preoperative, at implant, in the early postoperative period, at 1 year (between 11 and 13 months postoperatively), and annually for 8 years. The duration of the study is anticipated to be 8 years.

ELIGIBILITY:
Inclusion Criteria:

1. Patients is indicated for Mitroflow DL implantation according to the Instructions for Use (IFU).
2. Patient or patient's legal representative is willing to sign the informed consent.
3. Patient's preoperative evaluation indicated the need for native or prosthetic aortic valve replacement
4. Any patient amenable to aortic valve replacement with a biological prosthesis should be enrolled in the study, even in conjuction with valve repair, coronary artery bypass grafting and other procedures
5. Patient is able to return for all follow-up evaluations for the duration of the study (geographically stable).

Exclusion Criteria:

1. Patient is contra-indicated for Mitroflow DL implantation according to the Instructions for Use.
2. The patient has a pre-existing valve prosthesis in the mitral, pulmonary, or tricsupid position.
3. Patient requires a double or triple valve replacement (repair is not considered an exclusion).
4. Patient has active endocarditis or myocarditis.
5. Patient is pregnant or lactating.
6. Patient is participating in a concomitant research study of an investigational product.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of structural Valve Deterioration in Implanted Patients | 8 years
  To establish rates of structural valve deterioration through 8 years follow-up

SECONDARY OUTCOMES:
Early and Late Valve-Related Adverse Event Rates | Early (30 days) and Late (> 30 days)
  To determine early and late valve-related adverse event rates, including valve thrombosis, thromboembolism, paravalvular leak (all and major), bleeding(all and major), and endocarditis, for Mitroflow DL are comparable to appropriate historical controls
Early and Late Rates of hemolysis, non-structural valve dysfunction, valve-related embolism, re-operation, explant and death | Early (30 days) and Late (> 30 days)
  To determine rates of hemolysis, non-structural dysfunction, valve-related embolism, reoperation, explant and death (all cause and valve-related)
Hemodynamic Performance | 8 years
  To evaluate the hemodynamic performance of the Mitroflow DL valve as compared to other stented aortic bioprostheses in the current literature
Improvements in NYHA | 8 years
  To evaluate the overall improvements in patient condition by comparison of pre-operative and post-operative New York Heart Associate (NYHA) functional classification

CONTACTS AND LOCATIONS:
Overall Officials: John Kern, MD, Principal Investigator — University of Virginia
Locations (13):
- United States (13):
  - UCLA Medical Center, Los Angeles, California
  - Sharp Memorial Hospital, San Diego, California
  - River City Clinical Research, Jacksonville, Florida
  - UF Health - Jacksonville, Jacksonville, Florida
  - Watson Clinic Center for Research, Lakeland, Florida
  - Suburban Hospital - John Hopkins Medicine, Bethesda, Maryland
  - Bay Regional Medical Center, Bay City, Michigan
  - St. John Hospital & Medical Center, Detroit, Michigan
  - Catholic Medical Center, Manchester, New Hampshire
  - St. Joseph's Regional Medical Center, Paterson, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - University of Virginia Medical Center, Charlottesville, Virginia